CLINICAL TRIAL: NCT00702182
Title: Phase 1 Study of Oral Vinorelbine in Combination With Erlotinib in Advanced Non-Small Cell Lung Cancer (NSCLC) Using Two Different Schedules
Brief Title: Study of Oral Vinorelbine and Erlotinib in Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Principal Investigator, Wan-Teck Darren Lim, Senior Consultant, National Cancer Centre, Singapore
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPCTG-VEP1
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-10

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Lung Cancer; Vinorelbine; Erlotinib; Phase 1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Vinorelbine; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Vinorelbine, Erlotinib (Experimental): Escalating doses of vinorelbine on Day 1 and Day 8 of 21 Day cycle; Erlotinib 100 mg OD
  Interventions: Drug: Vinorelbine (Navelbine); Drug: Erlotinib
- Metronomic Vinorelbine, Erlotinib (Experimental): Escalating doses of vinorelbine TIW; erlotinib 100 mg OD
  Interventions: Drug: Vinorelbine (Navelbine); Drug: Erlotinib

INTERVENTIONS:
Drug: Vinorelbine (Navelbine) — Conventional Schedule Oral Vinorelbine on day 1 and day 8 of a 21 day schedule
  Other Names: Navelbine
  Arms: Conventional Vinorelbine, Erlotinib
Drug: Vinorelbine (Navelbine) — Metronomic Schedule Oral Vinorelbine 3 times a week
  Other Names: Navelbine
  Arms: Metronomic Vinorelbine, Erlotinib
Drug: Erlotinib — Daily Oral Erlotinib 100 mg
  Other Names: Tarceva

SUMMARY:
The purpose of this study is to define the schedule and dose of oral vinorelbine (Navelbine) to be used with erlotinib in non-small cell lung cancer.

DETAILED DESCRIPTION:
Additive or supraadditive activity of an EGFR TK-I with vinorelbine has been demonstrated in-vitro. Clinical synergism has also been described between gefitinib and vinorelbine in NSCLC. The use of cytotoxics in a metronomic schedule has not been well investigated in the clinical setting despite emerging pre-clinical data. Using an established oral cytotoxic such as oral vinorelbine in a metronomic dose-schedule is attractive due to the oral route of administration. Preclinical studies have shown that by using cytotoxics in a low-dose protracted manner, endothelial cells are preferentially affected via inhibition of proliferation and induction of apoptosis. In addition to this anti-angiogenic mechanism, an anti-vasculogenic process may also be involved that acts by reducing circulating endothelial progenitor mobilization and viability. Moreover, it has also been shown that tumours that were selected for high levels of acquired resistance to cytotoxics can be induced to respond by using metronomic doses of chemotherapy.

Continuous administration of metronomic oral vinorelbine, given three times a week, has been reported as feasible and well tolerated at doses up to 180 mg total dose per week. Early results showed activity against refractory solid tumors such as renal cancer, NSCLC, ovarian cancer, prostate cancer, unknown primary and Kaposi sarcoma.

This phase I study combines erlotinib and oral vinorelbine on two different schedules. The conventional schedule vinorelbine (CSV) aims to determine the MTD of conventional schedule of oral vinorelbine given on days 1 and 8 every 21 days plus daily erlotinib and the metronomic schedule vinorelbine (MSV) aims to determine the optimal metronomic dose of vinorelbine given 3 times a week plus daily erlotinib.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC
* At least one or two prior lines of chemotherapy for metastatic disease or locally advanced unresectable disease. There should be at least 4 weeks since prior chemotherapy or radiation therapy or 6 weeks if the last regimen included BCNU or mitomycin C
* Age > 21 years.
* ECOG performance status <2 (Karnofsky >60%, see Appendix A).
* Life expectancy of greater than 3 months
* Patients must have normal organ and marrow function as defined below:

  * leukocytes >3,000/mcL
  * absolute neutrophil count >1,500/mcL
  * platelets >100,000/mcL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) <2.5 X institutional ULN
  * creatinine within normal institutional limits OR
  * creatinine clearance >60 mL/min/1.73 m2
* The effects of Oral Vinorelbine on the developing human fetus are unknown. For this reason and because vinca alkaloids as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients may not be receiving any other investigational agents.
* Patients who have received previous vinorelbine or oral EGFR tyrosine kinase inhibitors
* Patients with progressive brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. However patients are eligible if they have brain metastases that have been treated with whole brain radiotherapy and are stable and not on corticosteroids.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Oral Vinorelbine or other agents used in study.
* Prior and / or concomitant treatment with drugs known to induce or inhibit cytochrome P450 3A4, CYP1A1 & CYP1A2 : phenytoin, carbamazepine, barbiturates, rifampicin, imidazole antifungals (such as ketoconazole, fluconazole, itraconazole, metronidazole), omeprazole and ritonavir
* Significant malabsorption syndrome or disease affecting the gastro-intestinal tract function
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnancy or breast feeding or women of child-bearing potential not using effective contraception,
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with Oral Vinorelbine. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* History of organ allograft
* Patients with evidence or history of bleeding diatheses or coagulopathy
* Serious, non-healing wound, ulcer, or bone fracture
* Because of interaction risk on CYP3A4, patients with concomitant treatments with vitamin K antagonists such as phenprocoumon or warfarin or heparin or heparinoids should be excluded

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-04; Primary Completion 2012-04 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Define the recommended dose of oral navelbine with erlotinib | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Teck Lim, MD, Principal Investigator — National Cancer Center Singapore
Locations (1):
- National Cancer Center Singapore, Singapore, Singapore

REFERENCES:
- [Derived] Sutiman N, Zhang Z, Tan EH, Ang MK, Tan SW, Toh CK, Ng QS, Chowbay B, Lim WT. Phase I Study of Oral Vinorelbine in Combination with Erlotinib in Advanced Non-Small Cell Lung Cancer (NSCLC) Using Two Different Schedules. PLoS One. 2016 May 2;11(5):e0154316. doi: 10.1371/journal.pone.0154316. eCollection 2016. PMID 27135612